# Exploration of Traumatic Brain Injury Clinical Trials: Unveiling Patient Participation Patterns

An Informed Consent Form For Power Clinical Trial's
Observational Study Involving Patients in Traumatic Brain Injury
Clinical Trials

Date: February 9, 2024

#### Introduction

Have you considered participating in a clinical trial for traumatic brain injury? Understanding why individuals choose to join, stay involved, or opt out of these trials is crucial for maximizing their impact. This invitation introduces you to our observational study seeking to answer this very question. Your participation, entirely voluntary and withdrawable at any time, holds significant value.

What does participating entail? Primarily completing questionnaires and participating in brief follow-up calls, designed to minimize any potential risks. While direct personal benefits may not be immediate, your contribution will fuel groundbreaking research to optimize clinical trial experiences for the traumatic brain injury community.

By uncovering the key factors influencing participation, we aim to develop more effective recruitment strategies and enhance patient engagement, ultimately leading to better treatment options and outcomes for individuals like you.

Before making your decision, we encourage you to thoroughly review the consent form and discuss any concerns with our research team, healthcare providers, or any trusted confidants. Remember, your informed choice is paramount.

#### Importance of Traumatic Brain Injury Clinical Trials

Clinical trials stand as cornerstones in the development of improved therapies for traumatic brain injury, yet concerns persist regarding the heterogeneity of participants. This study sheds light on the key factors influencing patient decisions to join, remain in, or rejoin traumatic brain injury clinical trials. Gaining insights into these motivations holds immense value for fostering more relevant and impactful research initiatives.

Our investigation prioritizes the recruitment of a diverse participant pool, enabling us to explore how aspects like age, ethnicity, socioeconomic status, and educational background influence participation choices. The data gathered will pave the way for crafting more effective strategies to engage underrepresented populations in future clinical trials.

Participation in this study is entirely voluntary, ensuring individuals can choose to withdraw at any time without repercussions. The study procedures, consisting mainly of completing questionnaires and follow-up calls, entail minimal risks. We strongly encourage potential participants to meticulously review the consent form and address any questions they may have.

Ultimately, this study strives to illuminate the underlying factors that shape participation in traumatic brain injury clinical trials. By boosting participation rates, we can accelerate the development of novel treatments for this debilitating condition.

## Exploring Factors That Shape Clinical Trial Participation

This observational study delves into the lived experiences of individuals with traumatic brain injury to understand their decision-making regarding clinical trial involvement. We aim to capture the nuances that influence their choices to join, remain in, or withdraw from these trials.

We seek individuals who participated in existing or completed interventional studies; both potential volunteers and participants identified through electronic medical records are welcome.

Upon expressing interest, participants receive a comprehensive informed consent form detailing the study's objectives and their rights. Data collection involves bi-weekly questionnaires exploring demographics, medical history, and factors influencing

participation. Additionally, in-depth, quarterly phone or video interviews will provide richer insights.

Statistical analysis of the data will identify key factors influencing patient participation. Our findings, shared through conferences and publications, will benefit all stakeholders involved in clinical trials.

This knowledge will directly impact future trials by informing the design, enhancing recruitment strategies, and improving retention rates, ultimately ensuring a more patient-centered research experience.

Participation is entirely voluntary, and withdrawal is possible at any stage without consequence. Completing surveys and participating in interviews pose minimal risk, with our readily available research team prepared to answer questions and address concerns promptly.

### Benefits of Traumatic Brain Injury Clinical Trials

Observational clinical trials for traumatic brain injury present a unique opportunity for patients to actively contribute to medical advancements and potentially enhance future treatment options.

Making an informed decision about participation requires careful consideration of individual circumstances and goals. Patients are encouraged to thoroughly evaluate potential benefits and risks, seeking guidance from their healthcare providers and the research team.

By participating in these trials, patients contribute valuable data that informs researchers about the natural progression of traumatic brain injury and the impact of existing treatments. This knowledge directly influences the development of more effective therapies, ultimately empowering patients to manage their condition with greater efficacy.

Joining an observational trial empowers individuals to become active participants in their healthcare journey, contributing to advancements that benefit not only themselves but also future generations of traumatic brain injury patients. Understanding Potential Risks in Traumatic Brain Injury Observational Studies

While observational studies of traumatic brain injury do not involve experimental treatments, there may be risks to consider before participation. These potential risks range from data privacy concerns to emotional distress related to the study topic and potential side effects from study procedures.

Prior to making a decision, it is crucial to meticulously review the informed consent document and openly discuss any questions or concerns with the research team. They are dedicated to providing clear and comprehensive information about potential risks, the study's benefits, and the safeguards in place to ensure participant safety and well-being.

Open communication is critical throughout the study. Should you feel uncomfortable or experience any adverse effects, you have the right to withdraw from participation at any time without penalty. Do not hesitate to voice your concerns to the research team, who are available to address them promptly and prioritize your welfare.

## **Factors Affecting Your Participation**

Clinical trials offer crucial avenues for medical advancements, but it's critical to recognize that your participation may end before the planned conclusion. Several factors beyond your direct control can lead to early termination, including study suspension, funding limitations, or concerns about your safety.

Additionally, factors within your control may also warrant termination, such as health changes, pregnancy, new information emerging during the trial, or inability to adhere to study procedures. Carefully considering these possibilities before enrolling is crucial for an informed decision about participation.

The informed consent process plays a significant role in understanding potential termination scenarios. Review the document thoroughly and discuss any concerns with the research team to ensure you fully comprehend the possibilities and your rights as a participant.

While early termination can be unexpected, remember that your agency remains protected. You have the right to withdraw at any time, with or without reason, and

without penalty. Open communication with the research team throughout the trial is encouraged to navigate any emerging concerns or questions.

## More Traumatic Brain Injury Clinical Trials

Taking part in clinical research for traumatic brain injury is entirely voluntary, and you have the complete freedom to withdraw without facing any consequences.

To gain a comprehensive understanding of ongoing traumatic brain injury research efforts, consider exploring Clinicaltrials.gov, a vast resource maintained by the National Institutes of Health (NIH). This platform houses information on numerous active studies around the world, allowing you to tailor your search based on your specific location and medical concerns.

Additionally, Power's reference page offers a regularly updated list of ongoing <u>traumatic</u> <u>brain injury clinical trials</u> currently seeking participants. Utilize these resources to explore various options and make informed decisions regarding your potential involvement.

Remember, participation is always voluntary, and your well-being remains the top priority. Take your time, carefully consider all available information, and don't hesitate to discuss your questions and concerns with healthcare professionals before making a decision.

## Online Resources at Your Fingertips

Seeking insightful explorations of clinical trial diversity? Look no further than the vast world of online resources. Here are two particularly valuable articles to consider:

Rutten-Jacobs, Loes, Tammy McIver, Adriana Reyes, Marta Pereira, Rachel Rosenthal, Christine T. Parusel, Kathryn R. Wagner, and Rachelle Doody. "Racial and ethnic diversity in global neuroscience clinical trials." *Contemporary Clinical Trials*Communications 37 (2024): 101255.

Liu, Jing Jing, Emma Davidson, and Aziz Sheikh. "Achieving ethnic diversity in trial recruitment." Pharmaceutical Medicine 25 (2011): 215-222.

These readily accessible resources dissect the intricacies of diversity in clinical trials, offering tangible strategies to promote inclusivity within research endeavors. Explore these articles and empower yourself to navigate the landscape of clinical research with a critical eye towards diversity and representation.

Prioritizing Your Privacy: Understanding Data Protections in This Research

We are firmly committed to safeguarding the privacy of your data throughout this research investigation. While absolute confidentiality cannot be guaranteed in every circumstance, we have implemented rigorous measures to ensure its protection. It's essential to understand that legal obligations may require the disclosure of personal information in certain situations.

However, we prioritize your anonymity in all research publications and presentations by omitting your name and any other personally identifiable details.

Access to your medical information for research, quality assurance, and data analysis purposes might be granted to select entities, such as accrediting bodies, government agencies (FDA, OHRP), safety monitors, study sponsors, and authorized representatives.

In specific instances, we may request your authorization for the use and sharing of your information within this study through an "Authorization Form." Your explicit consent will always be sought before sharing your information or research samples with Power researchers, other institutions, or external commercial entities for future research endeavors. Be assured that your confidential data will be handled securely and will be deleted appropriately when no longer needed.

## Participant's Consent

Signing this consent form signifies your acknowledgment and agreement to the following crucial aspects:

 You have meticulously reviewed and grasped the entirety of this informed consent form. We encourage you to seek diverse perspectives before making a decision, ensuring your choice is fully informed.

- All your questions concerning the research project and its methodology have been satisfactorily answered, empowering you with the necessary knowledge to participate confidently.
- You have carefully considered the potential benefits, risks, and alternative options associated with your involvement in the research.
- Your voluntary participation in this study does not compromise your legal rights in any way.
- We are committed to promptly communicating any significant updates that could impact your decision to continue participating in the research.
- You have the opportunity to raise any lingering questions or concerns before officially signing this consent form.

By understanding these critical points, you make a well-informed and responsible decision about your participation in this research endeavor.

| Participant's Signature | | |
|-------------------------|--------------------------|------|
| Name of Participant | Signature of Participant | Date |

Acknowledging Informed Consent: Ensuring Mutual Understanding

As the researcher, I have fulfilled my responsibility to engage in clear and comprehensive communication with the patient. All inquiries regarding the study, its methodology, and potential implications have been addressed to their satisfaction. Importantly, we have reaffirmed the voluntary nature of the patient's participation, ensuring their decision is fully informed and made with complete understanding.

By prioritizing open dialogue and respecting individual autonomy, we establish a foundation of trust and mutual respect essential for successful research collaboration.

| Signature of Researcher Who Rec | ceived Consent | |
|---------------------------------|---------------------------|------|
| Name of Investigator | Signature of Investigator | Date |